CLINICAL TRIAL: NCT02759874
Title: Prevention of Fetal Alcohol Spectrum Disorder (FASD) by the Use of Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Institute of Health Economics, Canada (Other)
Collaborators: University of Alberta (Other); SoberLink, LLC (Industry); Alberta Innovates Health Solutions (Other); Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00055644
Record Dates: First submitted 2016-04-28; First posted 2016-05-03 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Alcoholism; Pregnancy
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Intervention is pregnant women enrolled and using specialized breathalyzer device w face recognition technology linked to a cellphone
  Interventions: Device: specialized breathalyzer w face recognition technology
- Control Group (No Intervention): No intervention. No breathalyzer given. Access granted by participant to IHE to collect data from Alberta Health Services (medical records)

INTERVENTIONS:
Device: specialized breathalyzer w face recognition technology
  Other Names: Soberlink
  Arms: Experimental

SUMMARY:
The Institute of Health Economics is conducting a study to determine how a breathalyzer linked to a cloud based alcohol monitoring system changes alcohol consumption during pregnancy in women with alcohol dependency issues.

IHE posits that the ability to self-monitor blood alcohol concentration and the ability to share sobriety via email or text with loved ones and counselors may reduce alcohol consumption and thus reduce the possibility of delivering a child with FASD.

The study will provide useful evidence for tailoring future optimal maternal and child healthcare for women, with the potential of decreasing healthcare utilization by prevention of FASD. Breathalyzer device usage plus secure document sobriety should improve patient monitoring convenience and demonstrate reductions in alcohol use outside of traditional office visits and patient self-reports.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, Alcoholic, actively in treatment for alcoholism addiction

Exclusion Criteria:

* Not pregnant, not in treatment/therapy for addiction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Change in FASD Birthrate Levels | 3 years
  Binary- yes or no dx FASD within 3 years of birth

CONTACTS AND LOCATIONS:
Overall Officials: Andy Greenshaw, PhD, Principal Investigator — Department of Psychiatry, University of Alberta; Egon Jonsson, PhD, Study Director — Institute of Health Economics Executive Director and CEO